CLINICAL TRIAL: NCT04787705
Title: Novel Model of Preoperative Predictors of Outcome for Adults Undergoing Congenital Cardiac Surgery: Multicenter Model Validation
Brief Title: Multicenter Validation of a Predictor Model of ACHD Patients and Cardiac Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Providence Healthcare (Other); Montreal Heart Institute (Other); Auckland City Hospital (Other Government); Melbourne Health (Other)
Responsible Party: Sponsor
Other Study IDs: 18-5588
Record Dates: First submitted 2021-03-02; First posted 2021-03-09 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Adult Congenital Heart Disease; Cardiac Surgery
Keywords: Prediction model
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This multicentre study is to validate prediction modeling for the ACHD population undergoing cardiac surgery. The validation of this prediction model will support and generalize its use as a risk stratification tool in the ACHD population.

DETAILED DESCRIPTION:
The prediction model resulted from a preceding study, which uniquely based on comorbidities, was developed using 783 adults (>16 years) who underwent surgery for congenital heart disease at Toronto General Hospital (TGH) during 2004-2015. It identifies five pre-operative variables, namely presence of cognitive impairment, hepatic function, >3 chest incisions, anatomy diagnosis, and Body Mass Index <20 and >28, as significant predictors of composite adverse outcomes such as in-hospital mortality, prolonged ventilation (exceeding 7 days) and acute kidney injury.

This newly prediction model developed in a single-center has only been internally validated. It requires further external validation to demonstrate its utility in ACHD populations who require cardiac surgery in other cardiac institutions both nationally and internationally.

ELIGIBILITY:
Inclusion Criteria:

* all ACHD patients >16 years of age undergoing cardiac surgery requiring an open sternotomy or thoracotomy and cardiopulmonary bypass (CPB) or CPB standby at TGH and the collaborating institutions from April 2019.

Exclusion Criteria:

* CHD patients <16 years of age
* ACHD patients undergoing chest wall debridement and chest re-explorations for bleeding
* Non-cardiac surgery procedures and cardiology laboratory interventions

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All ACHD patients undergoing cardiac surgery in TGH and the other collaborating cardiac centers.
Sampling Method: Non-Probability Sample
Enrollment: 547 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Composite adverse events | 30 days from the day of surgery.
  The composite adverse outcome is defined by in-hospital mortality, prolonged ventilation (exceeding seven days), or acute kidney injury requiring dialysis.

SECONDARY OUTCOMES:
One-year mortality | 365 days from the day of surgery.
  One-year is defined as 365 days from the day of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Heggie, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital - University Health Network, Toronto, Ontario, Canada